CLINICAL TRIAL: NCT05596422
Title: Understand the Outcomes of Inflammatory Bowel Disease (IBD) Patients Treated With Biologics in Taiwan - A Decentralized Vedolizumab and Biologic Agents Core Assessments in IBD Collaboration
Brief Title: A Study of Vedolizumab and Biologic Agents in Participants With Inflammatory Bowel Disease (IBD)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4030
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Disease (IBD); Ulcerative Colitis; Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants With Biologics Discontinuation: Participants with IBD (UC or CD) who had received biologic treatments for at least 6 months after the initial confirmed diagnosis of IBD, and with at least 3 months follow-up period after biologics discontinuation will be observed retrospectively.
- Cohort 2: Participants Treated With Biologics: Participants with IBD (UC or CD) who had any dose of biologic for IBD treatment after the initial confirmed diagnosis of IBD will be observed retrospectively.

SUMMARY:
This is a non-interventional, retrospective study of adult participants with IBD. IBD consists of either ulcerative colitis (UC) or Crohn's disease (CD). The study will review the clinical data previously collected during February 2007 to March 2020 of approximately 724 participants who have had treatment with adalimumab, infliximab, golimumab, or vedolizumab in Taiwan.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective study in newly diagnosed IBD participants (UC or CD) treated with biologics.

The study will assess IBD relapse, effectiveness, and safety of biologic treatments in IBD participants. The study will enroll approximately 724 participants. The data will be collected from the electronic medical record (EMR) database of selected medical centers in Taiwan. IBD Participants who were evaluated and treated at the participating sites between 01 February 2007 to 31 March 2020 will be included. Participants will be assigned to the following two observational cohorts based on pathological diagnosis:

* Cohort 1: Participants With Biologics Discontinuation
* Cohort 2: Participants Treated With Biologics

This multi-center trial will be conducted in Taiwan. The overall duration of the study will be approximately 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed during February 2008 to March 2020 (or per local institutional review board [IRB] permitted date).

   * CD (International Classification of Diseases, Ninth Revision, Clinical Modification [ICD-9-CM]: 555.X or International Classification of Diseases, Tenth Revision, Clinical Modification [ICD-10-CM]: K50.XX, K50.XXX)
   * UC (ICD-9-CM: 556.X or ICD-10-CM: K51.XX, K51.XXX).
2. Had received any dose of biologics for IBD treatment, including vedolizumab adalimumab, infliximab or golimumab, from February 2008 to March 2020 (or per local IRB permitted date).

Exclusion Criteria:

1. Participants with any suspected diagnosis of CD or UC within one year before the initial date of confirmed IBD diagnosis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed IBD participants treated with biologics including vedolizumab, adalimumab, infliximab, or golimumab will be included in this study.
Sampling Method: Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Had IBD Relapse | Up to approximately 13 years
  IBD Relapse includes re-treatment with biologics, steroid use, IBD-related hospitalization record, IBD-related ER visits, IBD-related surgery, increase in disease index. The occurrence of any of the above records will be regarded as an IBD relapse.
Time to Relapse After Biologics Discontinuation | Up to approximately 13 years
  Time to relapse is defined as the time interval from end of treatment (EOT) to the first IBD relapse.
Correlation Between the Clinical Variables and Relapse Post Biologics Discontinuation | Up to approximately 13 years
  The identifying predictors of relapse, survival distributions will be studied using the log-rank test for the univariate analysis and then using time dependent Cox regression models for the multivariate analysis. The potential confounders of relapse including demographics, disease status, IBD-related treatment, symptom control treatment, lab and complication will be assessed. Two predictive models will be built in the study, one is "on biologics treatment", and other is "off biologics treatment".
Percentage of Participants Achieving Clinical Response | Up to approximately 13 years
  Clinical Response for CD is defined as Crohn's disease active index (CDAI) greater than or equal to (>=) 70 points reduction from the index date. For UC, Mayo score >=3 points reduction and >=30 percent (%) decrease from the index date with an accompanying rectal bleeding subscore >=1 points reduction or with absolute rectal bleeding subscore less than or equal to (<=) 1 and as >=2 point reduction in partial Mayo score. Index date: date when the first dose of the biologic was prescribed in each treatment cycle.
Percentage of Participants Achieving Clinical Remission | Up to approximately 13 years
  Clinical Remission for CD is defined as CDAI <=150 point.CDAI assesses CD based on clinical signs such as number of liquid stools,intensity of abdominal pain,general wellbeing,presence of comorbid conditions,antidiarrheal use,physical examination and laboratory findings.Total score ranges from 0 to 600 points.Clinical Remission for UC is defined as Mayo score <=2 and no individual subscore >1 and partial Mayo score <=1.Mayo score measure disease activity of UC.Mayo score consists of 4 sub-scores: stool pattern,most severe rectal bleeding of the day,endoscopic findings,global assessment by physician,each graded from 0 to 3 with higher scores indicating more severe disease.Scores are summed to give a total score range of 0 to 12.Partial Mayo score consists of 3 sub-scores:stool pattern,most severe rectal bleeding of the day, global assessment by physician, each graded from 0 to 3 with higher scores indicating more severe disease.Scores are summed to give a total score range of 0 to 9.
Percentage of Participants Achieving Steroid-free Remission | Up to approximately 13 years
  Steroid-free remission for CD is defined as CDAI <=150 point. CDAI assesses CD based on clinical signs such as number of liquid stools, intensity of abdominal pain, general wellbeing, presence of comorbid conditions, antidiarrheal use, physical examination and laboratory findings. Total score ranges from 0 to 600 points. Steroid-free remission for UC is defined as absence of steroid treatment (within 1 week before and after the date of potential clinical remission achieved) among participants on steroids at baseline (index date). Index date: date when the first dose of the biologic was prescribed in each treatment cycle.
Percentage of Participants Achieving Mucosal Healing | Up to approximately 13 years
  Mucosal healing is defined as absence of any symptom finding of ulcer or spontaneous bleeding on endoscopic assessment or Crohn's Disease Endoscopic Index of Severity (CDEIS) less than (<) 4 for CD participants and as Mayo endoscopic subscore <=1 for UC participants.
Correlation Between the Clinical Variables and Treatment Effectiveness | Up to approximately 13 years
  The relationship between clinical variables and treatment effectiveness will be assessed. The impact of potential bias from the baseline/demographic variables, baseline matching will be performed using propensity score 1:1 matching by each treatment cycle and different types of biologic treatments before performing the comparative analysis for effectiveness outcome. The matching condition will be determined according to the data collection. IBD participants with clinical response, clinical remission, steroid-free remission, and mucosal healing will be analyzed. The difference in effectiveness between IBD participants receiving different types of biologic treatment will be compared using Chi-square test.
Percentage of Participants Experiencing Infection | Up to approximately 13 years
  Participants experiencing opportunistic infections, hepatic viral infections, gastrointestinal (GI) infections, respiratory infections, respiratory failure, or sepsis or septic shock among participants receiving vedolizumab versus those receiving anti-TNF-α will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/d26e9d1a72ba4727?idFilter=%5B%22Vedolizumab-4030%22%5D